CLINICAL TRIAL: NCT06824779
Title: Impact of Influenza Vaccination on Nasal Resident Memory Immune Responses and Peripheral Respiratory-tropic Memory Immune Responses
Brief Title: Impact of FLU Vaccination on Nasal Resident Memory Immune Responses and Peripheral Respiratory-tropic Memory Immune Responses
Acronym: MUCOVAC_2
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24CH249; 2025-521217-46-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-16; First posted 2025-02-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Volunteers; Flu Vaccine
Keywords: Flu Vaccine; Nasal immune cells; airway immunity; memory immune responses
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLU VACCINATION (Experimental): Flu vaccination by one of FLU vaccines in the french market : FluarixTetra® (GSK), VaxigripTetra® (Sanofi-Pasteur), Influvac Tetra® (VIATRIS MEDICAL)
  Interventions: Drug: Flu Vaccine; Biological: Biological samples

INTERVENTIONS:
Drug: Flu Vaccine — Vaccination against FLU by one of FLU vaccines in the french market
Biological: Biological samples — Before and after the FLU vaccination, according the french recommendations, the following samples will be collected :
  Nasal fluid sampling Saliva sampling Blood samples Nasal cell sampling

SUMMARY:
Mucosal sites, such as respiratory mucosa, are the primary entry points entry points for pathogens. However, clinical evaluation of vaccines against respiratory respiratory pathogens is currently based primarily on analysis of systemic, i.e. peripheral antibody and cellular responses. These measurements give little indication of the immune responses in respiratory tissues tissues, even though the latter are essential for protection against infection. Protective immune responses in mucous membranes, including respiratory including respiratory tissues, rely on secretory IgA to neutralize pathogens neutralization of pathogens on the mucosal surface, as well as the development of the development of cellular responses, notably those from T (Trm) and B (Brm) lymphocytes. Preclinical studies and a few human studies have demonstrated that Trm are a crucial element mucosal protection against viral and bacterial infections. In fact it has been shown that resident memory lymphocytes, including Trm, are able to able to reside in nasal, pulmonary, intestinal, genital and skin mucosa and skin after infection.

DETAILED DESCRIPTION:
An initial MUCOVAC clinical trial (NCT06469359), sponsored by the CHU of Saint-Etienne and in collaboration with Jean Monnet University (GROUPE ON MUCOSAL IMMUNITY AND PATHOGENS (GIMAP)) has made it possible to set up a methodology for collecting and analysis of nasal resident memory T and B lymphocytes, and to detect peripheral memory lymphocytes that have the capacity to migrate into respiratory tissues. In this randomized cross-over study, the investigators investigators compared three nasal cell harvesting devices in a cohort of a cohort of healthy volunteers: (i) a nylon swab (FlowSwab, Copan Diagnostics), (ii) a plastic curette (Rhino-pro curette, Arlington Scientifc) and (iii) a mini cytological brush (Microm Microtech). This study determined that the nylon swab (data not yet published) is the most to collect viable memory resident lymphocytes from the nasal sphere.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to the Social Security System
* Signed informed consent form
* Having decided to be vaccinated against the flu

Exclusion Criteria:

* History of recurrent nosebleeds or systemic hemorrhages
* Previous injury or surgery which modified nasal cavity (e.g. deviated nasal septum)
* Individuals receiving anticoagulant therapy
* Individuals who experienced a severe respiratory infection leading to hospitalization in the last 6 months
* Individuals who received an antibiotic therapy for respiratory infection or any other infection in the last 6 months
* Immunocompromised individuals, or individuals taking immunosuppressed therapy or having a pathology (chronic infection, auto-immune disease) which could impact on immunity based on investigator's opinion
* Allergy to any component of the vaccines used in the study
* Unstable chronic pathology
* People deprived of liberty or hospitalized without any consent
* People under guardianship (authorship or curators)
* Individuals who received a vaccine (any vaccine) in the last 30 days
* Pregnant or breast-feeding people
* Individuals experiencing respiratory infection symptoms. Inclusion will be postponed up to 7 days after the symptom resolution
* People with no command of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-12-05 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of resident memory lymphocytes in the nasal mucosa measured by FLOQSwab | one month post vaccination

SECONDARY OUTCOMES:
Frequencies of resident memory T and B lymphocytes | one month post vaccination
Expression levels of respiratory mucosal migration markers on peripheral memory lymphocytes | one month post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane PAUL, PhD, Study Director — CHU de Saint-Etienne; Stéphanie LONGUET, PhD, Study Chair — Université de Saint-Etienne; Elisabeth BOTELHO-NEVERS, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No